CLINICAL TRIAL: NCT01989884
Title: Multicenter, Single Arm, Open-Label Phase II Trial On The Efficacy Of Ortataxel In Recurrent Glioblastoma
Brief Title: An Efficacy Study Of Ortataxel In Recurrent Glioblastoma
Acronym: Ortataxel
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRFMN-GBM-6272
Record Dates: First submitted 2013-10-23; First posted 2013-11-21 (Estimated); Last update posted 2019-10-23 (Actual); Status verified 2014-11

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — IDN 5109

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ortataxel (Experimental): 75 on day 1 every 21 days mg/m2 milligram(s)/square meter (intravenous use)
  Interventions: Drug: Ortataxel

INTERVENTIONS:
Drug: Ortataxel — 75 mg/m2, IV (in the vein) every 21 days. Number of Cycles: until progression or unacceptable toxicity develops.
  Other Names: IDN5109

SUMMARY:
Italian Study On The Efficacy Of Ortataxel In Recurrent Glioblastoma

DETAILED DESCRIPTION:
In this phase II study, adult patients with histologically confirmed GBM in recurrence after surgery or biopsy, standard radiotherapy and chemotherapy with temozolomide were eligible. Patients included were treated with ortataxel 75 mg/m² i.v. every 3 weeks until disease progression. The primary objective of the study was to evaluate the efficacy of ortataxel in terms of progression free survival at six months after the enrolment (PFS-6).

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed GBM.
* GBM in recurrence/progression after surgery (or biopsy), standard radiotherapy and chemotherapy with Temozolomide.
* Imaging confirmation of first tumor progression or regrowth as defined by the RANO criteria.
* No more than one prior line of chemotherapy (Temozolomide).
* Recovery from the toxic effects of prior therapy.
* Patients who have undergone recent surgery for recurrent or progressive tumor are eligible provided that:

  1. Surgery must have confirmed the recurrence.
  2. A minimum of 14 days must have elapsed from the day of surgery to registration. For core or needle biopsy, a minimum of 7 days must have elapsed prior to registration.
  3. Craniotomy or intracranial biopsy site must be adequately healed and free of drainage or cellulitis, and the underlying cranioplasty must appear intact at the time of registration.
* Age ≥ 18 years.
* Willingness and ability to provide written informed consent and to comply with the study protocol as judged by the investigator.
* Karnofsky-PS ≥ 60%.
* Stable or decreasing dose of corticosteroids within 5 days prior to registration.

Exclusion Criteria:

* Patients unable to undergo brain MRI scans with gadolinium (iv).
* Pre-existing peripheral neuropathy, grade ≥ 2.
* History of intracranial abscess within 6 months prior to registration.
* Anticipation of need for major surgical procedure during the course of the trial.
* Treatment with enzyme inducing antiepileptic agents was not allowed. However, patients whose anticonvulsant was changed to a nonenzymeinducing antiepileptic drug were eligible for entry after a 1-week ''washout'' period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2013-11; Primary Completion 2015-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
progression free survival-6 | after 6 months after randomization
  defined as the percentage of patients who are alive and progression free at 6 months after the randomization

SECONDARY OUTCOMES:
progression free survival | after 9 months of follow-up for each patient
  defined for each patient as the time from the date of randomization to the date of first progression, second primary malignancy or death from any cause, whichever comes first. Subjects not progressed or died at the time of the analysis will be censored at the last disease assessment date
Overall survival-9 | 9 months after randomization
  defined as the percentage of patients who are alive at 9 months after the randomization.
Objective response rate | after 9 months of follow-up for each patient
  defined as the percentage of patients who are judged by the Investigators to have an objective response as determined by the RANO criteria
Number of patients with AEs, SAEs, SADRs, SUSARs | after 9 months of follow-up for each patient
  * Incidence, nature, severity and seriousness of AEs, according of National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 4.0
  * Maximum toxicity grade experienced by each patient for each specific toxicity
  * Percentage of patients experiencing grade 3-4 toxicity for each specific toxicity
  * Patients with at least a SAE
  * Patients with at least a serious adverse drug reaction (SADR)
  * Patients with at least a suspect unexpected serious adverse reaction (SUSAR).
treatment compliance | 9 months after randomization
  -Dose-intensity, -percentage of patients with dose and/or time modifications, - Percentage of premature withdrawals

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Silvani, MD, Principal Investigator — Fondazione IRCCS Istituto Neurologico "Carlo Besta" di Milano
Locations (7):
- Italy (7):
  - Ospedale di Lecco, Lecco
  - Carlo Besta Neurological Foundation, Milan
  - A.O. OSpedale Niguarda Ca' Granda, Milan
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - Fondazione "Salvatore Maugeri", Pavia
  - IRCCS Fondazione "Casimiro Mondino", Pavia
  - Istituti Fisioterapici Ospitalieri, Rome

REFERENCES:
- [Result] Silvani A, De Simone I, Fregoni V, Biagioli E, Marchioni E, Caroli M, Salmaggi A, Pace A, Torri V, Gaviani P, Quaquarini E, Simonetti G, Rulli E, D'Incalci M; Italian Association of Neuro-Oncology. Multicenter, single arm, phase II trial on the efficacy of ortataxel in recurrent glioblastoma. J Neurooncol. 2019 May;142(3):455-462. doi: 10.1007/s11060-019-03116-z. Epub 2019 Feb 6. PMID 30726533
- See also: journal article — https://doi.org/10.1007/s11060-019-03116-z
- Available data/document: Clinical Study Report — https://doi.org/10.1007/s11060-019-03116-z